CLINICAL TRIAL: NCT03727477
Title: Efficacy of Treatment Sequences in Patients With ALK and ROS-1 Positive Non-small Cell Lung Cancer Who Received Lorlatinib as Part of the French Expanded Access Program
Brief Title: Efficacy of Treatment Sequences in Patients With Non-small Cell Lung Cancer Receiving Lorlatinib
Acronym: LORLATU
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: IFCT-1803
Record Dates: First submitted 2018-10-29; First posted 2018-11-01 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Non-small Cell Lung Cancer Metastatic; ALK Gene Rearrangement Positive; ROS-1 Gene Rearrangement Positive
Keywords: lorlatinib; Non-small Cell Lung Cancer; IFCT; Real-world study
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will evaluate progression-free survival, overall survival, best response and duration of treatment in patients with advanced ALK- and ROS1-positive non-small cell lung cancer who received lorlatinib as part of the French expanded access program.

DETAILED DESCRIPTION:
IFCT-1803 LORLATU study will evaluate progression-free survival, overall survival, best response and duration of treatment in patients with advanced ALK- and ROS1-positive non-small cell lung cancer who received lorlatinib (PF-06463922) as part of the French expanded access program. Those outcomes will be correlated to clinical, pathological, and radiological characteristics of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed locally advanced or metastatic NSCLC (Stage IIIB or IV accordingly to American Joint Committee on Cancer [AJCC] classification) at time of lorlatinib initiation
* Patients who received at least one week of treatment with lorlatinib as part of the French Expanded Access Program (ATU program); ATU was granted due to their inability to meet eligibility criteria for on-going recruiting trials, inability to participate in other clinical trials (e.g., poor performance status, lack of geographic proximity), or because other medical interventions are not considered appropriate or acceptable.

Exclusion Criteria:

* Patients enrolled in a lorlatinib clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed locally advanced or metastatic NSCLC who received at least one week of treatment with lorlatinib as part of the French Expanded Access Program (ATU program).
  Selection period would start at October 2015 (e.g.,initiation of lorlatinib treatment)
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | October 2015 - December 2019
  time from first dose of treatment to first occurrence of disease progression or death from any cause during the study

SECONDARY OUTCOMES:
Best response | October 2015 - December 2019
  best response recorded from the start of treatment until disease progression or start of further anti-cancer treatment
Duration of treatment | October 2015 - December 2019
  time from first dose of treatment to discontinuation of treatment or death from any cause during the study
Pattern of tumor progression | October 2015 - December 2019
  site of disease progression after each line of treatment
Reason for treatment discontinuation | October 2015 - December 2019
  this may be disease progression, toxicity, death, other
Duration of treatment beyond progression | October 2015 - December 2019
  time between first occurrence of disease progression and discontinuation the treatment
Central Nervous System (CNS) best response | October 2015 - December 2019
  in patients with CNS measurable lesion, best response on CNS locations recorded from the start of treatment until disease progression or start of further anti-cancer treatment
Central Nervous System (CNS) Progression free survival | October 2015 - December 2019
  time from first dose of treatment to first occurrence of disease progression in the CNS or death from any cause during the study
Overall Survival | October 2015 - December 2019
  is defined as the time from the first dose of treatment dose and death from any cause
Adverse Events | October 2015 - December 2019
  complications of lorlatinib therapy will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Girard, MD, PhD, Principal Investigator — Institut Curie Paris
Locations (30):
- France (30):
  - Aix-en-Provence - CH, Aix-en-Provence
  - Angers - CHU, Angers
  - Annemasse - CH, Annemasse
  - Avignon - CH, Avignon
  - Bordeaux - Polyclinique, Bordeaux
  - Brest - Morvan CHU, Brest
  - Cahors - CH, Cahors
  - Chartres-CH, Chartres
  - Clermont-Ferrand - CHU, Clermont-Ferrand
  - Colmar - CH, Colmar
  - Créteil - CHI, Créteil
  - La Roche-Sur-Yon - CH, La Roche-sur-Yon
  - Libourne - CH, Libourne
  - Lorient - CHBS, Lorient
  - Lyon - CRLCC, Lyon
  - Marseille - CRLCC, Marseille
  - Montpellier - ICM, Montpellier
  - Mulhouse - GHRMSA, Mulhouse
  - Paris - Curie, Paris
  - Paris - Saint-Louis, Paris
  - Paris - Tenon, Paris
  - Lyon - URCOT, Pierre-Bénite
  - Reims - CHU, Reims
  - Saint-Etienne - CHU, Saint-Etienne
  - Saint-Nazaire - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Toulouse - CHU, Toulouse
  - Tours - CHU, Tours
  - Valenciennes - Clinique, Valenciennes
  - Vandoeuvre-lès-Nancy - CRLCC, Vandœuvre-lès-Nancy
  - Villejuif - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Girard N, Galland-Girodet S, Avrillon V, Besse B, Duruisseaux M, Cadranel J, Otto J, Prevost A, Roch B, Bennouna J, Bouledrak K, Coudurier M, Egenod T, Lamy R, Ricordel C, Moro-Sibilot D, Odier L, Tillon-Strozyk J, Zalcman G, Missy P, Westeel V, Baldacci S. Lorlatinib for advanced ROS1+ non-small-cell lung cancer: results of the IFCT-1803 LORLATU study. ESMO Open. 2022 Apr;7(2):100418. doi: 10.1016/j.esmoop.2022.100418. Epub 2022 Feb 26. PMID 35227966
- [Result] Baldacci S, Besse B, Avrillon V, Mennecier B, Mazieres J, Dubray-Longeras P, Cortot AB, Descourt R, Doubre H, Quantin X, Duruisseaux M, Monnet I, Moro-Sibilot D, Cadranel J, Clement-Duchene C, Cousin S, Ricordel C, Merle P, Otto J, Schneider S, Langlais A, Morin F, Westeel V, Girard N. Lorlatinib for advanced anaplastic lymphoma kinase-positive non-small cell lung cancer: Results of the IFCT-1803 LORLATU cohort. Eur J Cancer. 2022 May;166:51-59. doi: 10.1016/j.ejca.2022.01.018. Epub 2022 Mar 9. PMID 35278825